CLINICAL TRIAL: NCT05006898
Title: Synergistic Use of Pilocarpine-Brimonidine-Oxymetazoline to Control Presbyopia Symptoms
Brief Title: Compound to Control Presbyopia Symptoms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Optall Vision (Other)
Responsible Party: Principal Investigator, Cesar Alejandro Sanchez Galeana, Principal Investigator, Optall Vision
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBOPC01
Record Dates: First submitted 2021-06-09; First posted 2021-08-16 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Pilocarpine; Brimonidine Tartrate; Oxymetazoline

STUDY DESIGN:
Intervention Model Description: Pilocarpine, brimonidine, oxymetazoline (PBO) compound was instilled in the non-dominant eye of presbyopic patients, while in the dominant eye pilocarpine or brimonidine were instilled.
Who Masked: Participant, Care Provider
Masking Description: While in office the care provider took a number out of a closed container. Number 1 was designated for the placebo; Number 2 was designated for the compound
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PBO Investigational drug (Experimental): Pilocarpine, brimonidine, oxymetazoline combined with hyaluronic acid and bromfenac combined in an ophthalmic solution to be randomly instilled in one eye.
  Interventions: Combination Product: PBO to control presbyopia symptoms
- Pilocarpine (Active Comparator): Pilocarpine was instilled in the other oye.
  Interventions: Combination Product: PBO to control presbyopia symptoms
- Brimonidine (Active Comparator): Brimonidine was instilled in the other eye.
  Interventions: Combination Product: PBO to control presbyopia symptoms

INTERVENTIONS:
Combination Product: PBO to control presbyopia symptoms — Low dose PBO to control presbyopia symptoms
  Other Names: Pilocarpine; Brimonidine; Oxymetazoline

SUMMARY:
Low dose compose to control presbyopia symptoms

DETAILED DESCRIPTION:
A los dose compound including pilocarpine, brimonidine and oxymetazoline was use to control presbyopia symptoms compared to pilocarpine and brimonidine in low doses.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* Presbyopic
* 40 - 59 years

Exclusion Criteria:

* Diabetics
* Previous eye surgery
* Previous eye disease
* > 0.50 myopia
* > 1.5 hyperopia or astigmatism

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Jaeger notation near uncorrected visual acuity change | 1 hour
  Number of lines improved 1 hour after drug instillation
Comparison of PBO compound Jaeger notation improvement vs Pilocarpine or Brimonidine alone | 1 hour
  Number of lines improve comparing PBO compound vs Pilocarpine or Brimonidine

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Alejandro S Galeana, Principal Investigator — Optall Vision
Locations (1):
- Optall Vision, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No